CLINICAL TRIAL: NCT06334926
Title: Prediction of Survival in Colorectal Cancer Patients on the Basis of Body Mass Index and Lymph Node Yield - a Retrospective Single Center Cohort Analysis Over a Quarter of a Century
Brief Title: BMI and Lymph Node Count in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Klinikum Floridsdorf (Other)
Collaborators: Medical University of Vienna (Other); Klinik Favoriten (Other); Salzkammergut Klinikum Vöcklabruck (Network)
Responsible Party: Principal Investigator, Dr. Tamara Braunschmid, MD, Klinikum Floridsdorf
Other Study IDs: EK 18-002-VK
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: The Aim of This Study is to Determine the Influence of BMI and Lymph Node Status on OS in CRC Patients in the Long Term
Keywords: colorectal cancer, survival, prognostic factors, body mass index, obesity paradox, lymph node count
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colon cancer patients: Retrospective data analysis of the subgroup of patients suffering from colon carcinoma
  Interventions: Other: no intervention, retrospective data analysis
- Rectal cancer patients: Retrospective data analysis of the subgroup of patients suffering from rectal carcinoma
  Interventions: Other: no intervention, retrospective data analysis

INTERVENTIONS:
Other: no intervention, retrospective data analysis — not applicable, retrospective data analysis

SUMMARY:
Background and aim: Colorectal Cancer (CRC) is one of the most frequent cancer entities in the western world. It is known that obesity is one of the major risk factors for CRC. In contrast, mild obesity seems to have a positive effect on postoperative outcome, which is known as the "obesity paradox". Also, the number of resected lymph nodes (LN) during surgery is very important for correct staging. The aim of the present project is to evaluate the impact of BMI and LN-yield on long term overall survival (OS) of CRC patients treated with curative intent.

Methods: Patients treated for CRC between 1998 and 2011 at the Klinik Favoriten in Vienna, Austria were analyzed in this retrospective single-center cohort analysis concerning OS.

ELIGIBILITY:
Inclusion Criteria:

* colorectal carcinoma
* treated at the Klinik Favoriten between 1998 and 2011
* elective or acute surgical setting
* curative intent
* older than 18 years

Exclusion Criteria:

* other carcinoma (anal, metastases, ...)
* treated before 1998 or after 2011
* palliative intent
* younger than 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had surgery at the department of surgery at the Klinik Favoriten between 1998 and 2011 were analyzed. 1192 patients met the inclusion criteria were therefore pseudonymized and recorded in a newly developed database.
Sampling Method: Non-Probability Sample
Enrollment: 1192 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
overall survival | median follow up of 11.3 years
  The aim of the present project is to evaluate the impact of BMI and LN-yield on long term overall survival (OS) of CRC patients treated with curative intent.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Braunschmid, MD, Principal Investigator — Klinik Floridsdorf
Locations (1):
- Klinik Floridsdorf, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
All relevant data will be shared within a publication of the study. Detailled data are available upon request